CLINICAL TRIAL: NCT02201446
Title: Relationship Between Elevated Soluble Cluster of Differentiation 74 (CD74) and Severity of Experimental and Clinical ALI/ARDS.
Brief Title: The Role of Circulating Soluble CD74 in Acute Lung Injury
Status: Completed | Type: Observational
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Zhaofan Xia, President, Changhai Hospital
Other Study IDs: 20131224
Record Dates: First submitted 2014-07-24; First posted 2014-07-28 (Estimated); Results first posted 2016-12-15 (Estimated); Last update posted 2017-02-17 (Actual); Status verified 2017-01

CONDITIONS: Acute Lung Injury; Acute Respiratory Distress Syndrome
MeSH Terms: conditions — Acute Lung Injury; Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — ARDS patients and healthy volunteers
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- ARDS patients: Eighty-one patients were enrolled consecutively over a two-year time period (2014-2015) and identified as ARDS prospectively according to the Berlin definitions of the European Society of Intensive Care Medicine and American Thoracic Society on ARDS. Exclusion criteria were an age of less than 16 years, pregnancy, chronic obstructive pulmonary disease according to medical history and failure to obtain informed consent.
- Healthy volunteers: Fifty-eight healthy volunteers recruited from the general population who had no significant medical history and no medications were categorized as control patients.

SUMMARY:
Efforts to identify circulating factors that predict severity of acute lung injury/acute respiratory distress syndrome（ALI/ARDS） patients is unrevealing. The primary purpose of this study is to verify our hypothesis that soluble CD74 might be a potential novel ALI/ARDS biomarker.

DETAILED DESCRIPTION:
Acute lung injury (ALI) or acute respiratory distress syndrome (ARDS) is a devastating cause of morbidity and mortality characterized by alveolar epithelial and endothelial injury. Despite recent advances in pathogenetic mechanisms and therapy strategies of ALI, efforts to identify circulating factors that predict severity of ALI/ARDS patients have been unrevealing.

CD74 (also known as a major histocompatibility complex (MHC) class II invariant chain) is a type II transmembrane protein, recently found to be the high-affinity receptor of macrophage migration inhibitory factor (MIF). MIF promotes neutrophil accumulation in alveolar space via binding to CD74 expressed on the cell surface. Our previous study， consistent with others, has shown that MIF was highly expressed in acute lung injury (ALI). In addition, we also detected highly CD74 expression in lipopolysaccharide (LPS)-induced ALI mouse model. Recently, a circulating form of CD74 was discovered in autoimmune liver disease. Similarly, we investigated the existence of soluble form of CD74 in serum and bronchoalveolar lavage fluid (BALF) in ALI mouse model and burn or trauma related ALI patients. Based on these finds, we postulated that soluble CD74 might participate in regulating lung inflammation and be a potential novel ALI/ARDS biomarker.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of ALI/ARDS
* Informed consent was obtained from either the subjects themselves or from designated surrogates before enrollment in the study.

Exclusion Criteria:

* Patients who have chronic lung disease before enrollment.
* Patients who have severe organ dysfunction, autoimmune diseases and tumor.
* Women who are pregnant or breast-feeding.
* Patients who, in the opinion of the Investigator, have any other medical condition which renders the patient unable to complete the study or which would interfere with optimal participation in the study or produce significant risk to the patient.
* Patients participating in or planning to enroll in another clinical trial during the time of the study.

Ages: 16 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with and without ARDS were screened from Changhai Hospital. Patients were enrolled consecutively over a 2-year time period (2014-2015). All enrolled patients with ALI met the American-European Consensus Committee criteria.In addition, healthy individuals were recruited from the general population.
Sampling Method: Non-Probability Sample
Enrollment: 139 (Actual)
Dates: Start 2014-03; Primary Completion 2014-11 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zhaofan Xia, MD PhD, Study Director — Department of Burn Sugery, Changhai Hospital
Locations (1):
- Department of Burn and Trauma Sugery, Changhai Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wu G, Sun Y, Wang K, Chen Z, Wang X, Chang F, Li T, Feng P, Xia Z. Relationship between elevated soluble CD74 and severity of experimental and clinical ALI/ARDS. Sci Rep. 2016 Jul 22;6:30067. doi: 10.1038/srep30067. PMID 27444250

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ARDS Patients | Healthy Volunteers
Started | 81 | 58
Completed | 81 | 58
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ARDS Patients | Healthy Volunteers | Total
Number analyzed (Participants) | 81 | 58 | 139
Age, Continuous [Mean (Standard Deviation); unit: years] — The age of participant.
  years | 48.02 (16.05) | 39.52 (10.43) | 44.47 (14.58)
Gender [Count of Participants; unit: Participants]
  Female | 37 | 26 | 63
  Male | 44 | 32 | 76
Sequential Organ Failure Assessment(SOFA) [Mean (Standard Deviation); unit: Scores on a scale] — SOFA score ranges from 0 to 43. A higher values represent a worse outcome.
  Scores on a scale | 7.16 (3.70) | NA (NA) — Not collected for healthy volunteers | 7.16 (3.70)
Trauma [Number; unit: participants] | 35 | 0 | 35
Inhalation injury [Number; unit: participants] | 46 | 0 | 46
Diabetes mellitus [Number; unit: participants] | 8 | 0 | 8
Hypertension [Number; unit: participants] | 15 | 0 | 15
Kidney disease [Number; unit: participants] | 2 | 0 | 2
Respiratory disease [Number; unit: participants] | 2 | 0 | 2
Blood diseases [Number; unit: participants] | 0 | 0 | 0
Day1 tumor necrosis factor-α(TNF-α) [Mean (Inter-Quartile Range); unit: pg/ml] | 97.09 [92.32 to 100.82] | NA [NA to NA] — not collected for healthy volunteers | 97.09 [92.32 to 100.82]
Day1 interleukin-6 (IL-6) [Mean (Inter-Quartile Range); unit: pg/ml] | 101.63 [79.5 to 138.9] | NA [NA to NA] — not collected for healthy volunteers | 101.63 [79.5 to 138.9]
Day1 migration inhibitory factor (MIF) [Mean (Standard Deviation); unit: ng/ml] | 73.64 (23.27) | NA (NA) — not collected for healthy volunteers | 73.64 (23.27)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Receiving Mechanical Ventilation
Time Frame: up to 28 days
Population: not collected for healthy volunteers
Measure: Number; unit: participants
Arm/Group | ARDS Patients | Healthy Volunteers
Number analyzed (Participants) | 81 | 58
participants | 51 | NA — not collected for healthy volunteers

2. Primary Outcome: Fraction of Inspired Oxygen (FiO2)/Partial Arterial Oxygen Pressure (PO2)
Time Frame: up to 28 days
Population: not collected for healthy volunteers
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | ARDS Patients | Healthy Volunteers
Number analyzed (Participants) | 81 | 58
ratio | 2.1 (0.46) | NA (NA) — not collected for healthy volunteers

3. Primary Outcome: Acute Physiology and Chronic Health Evaluation (APACHE) II Scores
Description: APACHE II scores range from 0 to 71. A higher values represent a worse outcome.
Time Frame: up to 28 days
Population: not collected for healthy volunteers
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | ARDS Patients | Healthy Volunteers
Number analyzed (Participants) | 81 | 58
Scores on a scale | 14.35 (6.39) | NA (NA) — not collected for healthy volunteers

4. Primary Outcome: Serum Soluble Cluster of Differentiations 74 (sCD74)
Description: The concentration of sCD74 was determined using Elx800 (BioTek Instruments, Inc. VT), and normalization was based on concentration-response curves, using CD74 recombinant protein.
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | ARDS Patients | Healthy Volunteers
Number analyzed (Participants) | 81 | 58
ng/ml | 87.04 (31.53) | -14.77 (15.57)

5. Primary Outcome: Serum Soluble Cluster of Differentiations 74 (sCD74)
Description: as for outcome 4
Time Frame: Day 3
Population: Only 62 ARDS patients with Day 3 blood samples were analyzed.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | ARDS Patients | Healthy Volunteers
Number analyzed (Participants) | 62 | 58
ng/ml | 132.92 (40.40) | -14.78 (15.57)

6. Secondary Outcome: Length of Stay in the ICU
Time Frame: 1 year
Population: not collected for healthy volunteers
Measure: Mean (Inter-Quartile Range); unit: days
Arm/Group | ARDS Patients | Healthy Volunteers
Number analyzed (Participants) | 81 | 58
days | 23 [15 to 44] | NA [NA to NA] — not collected for healthy volunteers

7. Secondary Outcome: Length of Hospital Stay
Time Frame: 1 year
Measure: Mean (Inter-Quartile Range); unit: days
Arm/Group | ARDS Patients | Healthy Volunteers
Number analyzed (Participants) | 81 | 58
days | 36.94 [22 to 53] | NA [NA to NA] — not collected for healthy volunteers

8. Secondary Outcome: Days of Unassisted Ventilation
Time Frame: 1 year
Measure: Mean (Inter-Quartile Range); unit: days
Arm/Group | ARDS Patients | Healthy Volunteers
Number analyzed (Participants) | 81 | 58
days | 22 [8.5 to 28] | NA [NA to NA] — not collected for healthy volunteers

9. Secondary Outcome: Death
Time Frame: up to 28 days
Measure: Number; unit: participants
Arm/Group | ARDS Patients | Healthy Volunteers
Number analyzed (Participants) | 81 | 58
participants | 14 | 0

10. Secondary Outcome: TNF-α
Time Frame: Day 3
Population: Only 62 ARDS patients with Day 3 blood samples were analyzed
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | ARDS Patients | Healthy Volunteers
Number analyzed (Participants) | 62 | 58
pg/ml | 138.67 (64.26) | NA (NA) — not collected for healthy volunteers

11. Secondary Outcome: IL-6
Time Frame: Day 3
Population: Only 62 ARDS patients with Day 3 blood samples were analyzed
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | ARDS Patients | Healthy Volunteers
Number analyzed (Participants) | 62 | 58
pg/ml | 305.36 (177.14) | NA (NA) — not collected for healthy volunteers

12. Secondary Outcome: MIF
Time Frame: Day 3
Population: Only 62 ARDS patients with Day 3 blood samples were analyzed
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | ARDS Patients | Healthy Volunteers
Number analyzed (Participants) | 62 | 58
ng/ml | 129.27 (41.12) | NA (NA) — not collected for healthy volunteers

ADVERSE EVENTS:
Time Frame: 1 month
Arm/Group | ARDS Patients | Healthy Volunteers
Serious Adverse Events (participants affected / at risk) | 14/81 | 0/58
Other Adverse Events (participants affected / at risk) | 0/81 | 0/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ARDS Patients (N=81) | Healthy Volunteers (N=58)
Heart failure (Cardiac disorders) | 0 (0) | 0 (0)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0)
Renal inadequacy (Renal and urinary disorders) | 0 (0) | 0 (0)
Respiratory infection (Infections and infestations) | 0 (0) | 0 (0)
Death (Respiratory, thoracic and mediastinal disorders) | 14 (14) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ARDS Patients (N=81) | Healthy Volunteers (N=58)
Astriction or diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0)
Anxiety or depression (Nervous system disorders) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0)
Fever (General disorders) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No